CLINICAL TRIAL: NCT03219801
Title: Evaluation of Safety and Efficacy in Patients With Systemic Lupus Erythematosus by Transplantation of Umbilical Cord Derived Mesenchymal Stem Cells
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Systemic Lupus Erythematosus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17277787D-SLE
Record Dates: First submitted 2017-07-10; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesenchymal stem cells (Experimental): Selected SLE patients were randomly divided into treated group and control group. In the treated group, 100-300 million allogeneic human umbilical cord derived mesenchymal stem cells were infused intravenously for one SLE patient. The possible adverse events, including immediately after mesenchymal stem cells infusions, as well as the long-term safety profiles were observed.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — SLE patients in the treated group were given human umbilical cord derived mesenchymal stem cells by intravenous infusion and conventional therapy. There was only conventional treatment in the control group. All patients after treatment for 1, 3 and 6months were evaluated respectively the curative effect.

SUMMARY:
This study is to evaluate the safety and efficacy of human umbilical cord derived mesenchymal stem cells transplantation in systemic lupus erythematosus.

DETAILED DESCRIPTION:
To ensure that all patients of systemic lupus erythematosus (SLE) completed 6-months follow-up, twenty SLE patients ranging from 14 to 60 years old were enrolled in this trial. Participants matched with the inclusion criteria were allocated randomly into two groups:Human Umbilical Cord Derived Mesenchymal Stem Cells (hUC-MSCs) treated group and control group. Clinical trials are being increasingly established to investigate the therapeutic potential of these cells for SLE. The aim of the present study is to investigate safety and efficacy of vein infusion of allogeneic hUC-MSCs in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SLE(Systemic lupus erythematosus) from American College of Rheumatology(ACR) according to established criteria in 1997
2. Age from 14 to 60 years
3. No serious infection or acute hemorrhage
4. Left ventricular ejection fraction (LVEF)≥ 50%
5. Both transaminase and serum creatinine level are more than twice times the upper limit of normal
6. No acute infectious diseases.
7. Understanding and willingness to sign a written informed consent document.

Exclusion Criteria:

Patients with SLE have to be disqualified from this study if any of the following is applicable:

1. SLE(Systemic lupus erythematosus) with severe infection.
2. Severe heart attack, liver and kidney disease following serious complications
3. Patients with allergic constitution.
4. Pregnancy and breastfeeding women.
5. Accompanied by malignant tumors or other malignant disease
6. Patients as participant in the other clinical text
7. Patients with active tuberculosis, acute sever hepatitis or infectious period of diseases.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of Complement levels(C3 and C4) in peripheral blood | Post cell transplantation: 1, 3, 6 months
  The recovery of immunologic function is evaluated by complement levels (g/L) in peripheral blood.

SECONDARY OUTCOMES:
Erythrocyte sedimentation rate | Post cell transplantation: 1, 3, 6 months
  The change of inflammation is evaluated by erythrocyte sedimentation rate.
C-reactive protein | Post cell transplantation: 1, 3, 6 months
  C-reactive protein is an acute phase reactants. It can be moderately increased in in peripheral blood of SLE patients.
adverse reaction | Post cell transplantation: 1, 3, 6 months
  Adverse reaction includes temperature changes(℃), the change of blood pressure(mmHg) and allergic reaction.These measurements were associated with the safety of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — The First Hospital of Hebei Medical University; Qingchi Liu Liu, Doctor, Study Director — The First Hospital of Hebei Medical University; Quanhai Li, Doctor, Study Director — The First Hospital of Hebei Medical University; Xiaohui Jia, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Xianyun Wang, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Fan Zhang, Bachelor, Principal Investigator — The First Hospital of Hebei Medical University; Yang Shen, Master, Principal Investigator — The First Hospital of Hebei Medical University; Bing Ma, Master, Principal Investigator — The First Hospital of Hebei Medical University; Wanyi Yin, Master, Principal Investigator — The First Hospital of Hebei Medical University; Dan Zhao, Master, Principal Investigator — The First Hospital of Hebei Medical University; Bojian Sun, Master, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No